CLINICAL TRIAL: NCT07399886
Title: PlAnt Vs Animal Based Oral Nutritional Supplements: Patients' Opinions and Nutritional Outcomes: A Multicenter Pilot Feasibility Study
Brief Title: Plant-based Versus Animal-based Oral Nutritional Supplements
Acronym: PAVOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht UMC (Unknown); Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-17931; FreP-001-IEN (Other: Fresenius Kabi Deutschland GmbH)
Record Dates: First submitted 2025-12-18; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Risk of Malnutrition
Keywords: plant-based ONS; animal-based ONS; Risk of malnutrition; pilot feasibility; hospitalized patients; oral nutritional drinks; plant protein; sustainability; medical nutrition

STUDY DESIGN:
Intervention Model Description: Patients that would get the advice of a dietitian to use two bottles of ONS a day will be eligible. So this is just part of the usual care. The amount ONS they will use during the study is also part of the usual care. So only the type of ONS will be determined by the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-based ONS (Experimental): In this arm, patients who are advised, as part of usual care, to use at least two bottles of oral nutritional supplements (ONS) per day are randomized to the plant-based group. Participants receive plant-based ONS, with the daily amount prescribed by the dietitian according to usual care.
  Interventions: Dietary Supplement: Fresubin Plant-based drink vanilla©
- Animal-based ONS (Experimental): In this arm, patients who are advised, as part of usual care, to use at least two bottles of oral nutritional supplements (ONS) per day are randomized to the animal-based group. Participants receive animal-based ONS, with the daily amount prescribed by the dietitian according to usual care.
  Interventions: Dietary Supplement: Fresubin Yodrink raspberry©

INTERVENTIONS:
Dietary Supplement: Fresubin Plant-based drink vanilla© — Patients will receive plant-based oral nutritional supplements (ONS). The amount of bottles ONS a day, will be based on their nutritional intake versus requirements by a dietitian. This is usual care, only the sort of ONS differs from normal care.
  Arms: Plant-based ONS
Dietary Supplement: Fresubin Yodrink raspberry© — Patients will receive animal-based oral nutritional supplements (ONS). The amount of bottles ONS a day, will be based on their nutritional intake versus requirements by a dietitian. This is usual care, only the sort of ONS differs from normal care.
  Arms: Animal-based ONS

SUMMARY:
Background information:

Many people who are admitted to the hospital are at risk of malnutrition. In some patient groups, this can be as high as 40%. When someone is not eating enough, the dietitian often recommends oral nutritional supplements (ONS). These are energy- and protein-rich drinks that help patients get enough nutrition. They can reduce complications, lower the chance of being readmitted to the hospital, and help improve body weight and physical functioning.

In the Netherlands, the Ministry of Health and the Dutch Federation of University Medical Centers have signed the Green Deal "Working together on sustainable care." One of the goals is to make healthcare greener and climate-neutral by 2026. This also applies to medical and non-medical nutrition, including ONS.

Because of this, there is increasing attention on developing ONS that contain more plant-based proteins, which may be more sustainable.

What do will the investigators find out?

It is unknown how plant-based ONS work when patients use them for a longer period of time. For example:

* Do they help patients get enough energy and protein?
* What are the effects on physical and clinical outcomes? Before a large study with many patients is started, it is important to first test whether this type of research is feasible.

Feasibility in terms of

* Recruitment rate
* Drop-out rate
* Adherence to the ONS advice
* Study measurements (succesfull vs unsuccesfull measurements)

To answer these questions, a smaller pilot study will be conducted in which plant-based ONS will be compared to animal-based ONS.

What does this study look like?

Inclusion criteria:

Patients from the departments of medical oncology, lung diseases, cardiology, cardiothoracic surgery, and orthopedics at Maastricht UMC+ and Radboudumc. These are patients who are currently not eating enough.

These patients receive advice from the dietitian to take at least two bottles of ONS per day. If they want to participate in the study, they will be randomly assigned to one of two products:

* Animal-based (milk protein): Fresubin YoDrink Raspberry©
* Plant-based (soy protein): Fresubin Plant-Based Drink Vanilla©

Measurements will be performed at the start of the study and again after three months. In the meantime, the researcher will contact the patient twice by phone to ask how things are going.

DETAILED DESCRIPTION:
Measurements that are being performed:

* weight and height
* fat- and muscle mass with the BIA
* muscle thickness with the lumify ultrasound
* handgrip strength
* physical performance tests (SPPB, TUG)
* questionnaires (about quality of life, habitual physical activity, and nutritional status)
* 3-day food diary

This will be performed at the start and after three months. In the mean time the patients will register their real intake of the ONS in a logbook every day. The amount of the ONS that the patients will drink in the mean time depends on the amount that the dieititan advices (usual care).

After one month and after two months the researcher will contact the patient and ask if there are any changes in their food intake, their weight, the advice of the dietitian, what they think of the ONS, discuss the logbook and they can ask their questions about the study. After three months the measurements will be performed again. Besides, an interview will be conducted about their experiences and perspectives of the ONS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical patients with cancer and lung diseases, cardiology patients, patients with cardiothoracic surgery, and orthopaedic patients age ≥18 years, and treated at Radboudumc or Maastricht UMC+.
* Patients who have been advised at least 2 bottles of ONS daily based on a high risk of malnutrition (MUST≥2, PG-SGA-SF≥ 9) and/or by the dietitians expertise.
* Written informed consent (IC)

Exclusion Criteria:

* Patients who are or become dependent on tube or parenteral nutrition
* Patients where life-extending therapy is no longer possible
* Unable to follow up study instructions
* Lactose intolerance
* Soy allergy/intolerance
* Vegan diet
* Patients who have used ONS in the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a multicenter RNIT study, assessed by recruitment rate defined as the percentage of patients who participated versus total numer of eligible patients. | From enrollment to the end of the study (three months after inclusion)
  Recruitment rate, defined as the proportion of patients who participate relative to the total number of eligible patients who are approached for participation.
  The recruitment rate will be calculated as the number of included participants divided by the number of approached eligible patients and will be reported as a percentage.
Feasibility of a multicenter RNIT study, assessed by drop-out rate, percentage of participants who discontinue the study. | From enrollment to end of study (three months after inclusion)
  Drop-out rate is defined as the percentage of participants who discontinue the study, the timing of drop-out, and the reported reasons for drop-out.
Feasibility of a multicenter RNIT study, assessed by adherence to oral nutritional supplements (ONS). Percentage of the prescribed ONS intake that is acutally consumed over the study period. | From enrollment to the end of the study (three months after inclusion)
  Adherence feasibility will be assessed using a daily logbook in which participants record the amount of oral nutritional supplements (ONS) consumed each day relative to the prescribed amount. Adherence will be calculated as the percentage of the prescribed ONS intake that is actually consumed over the study period.
Feasibility of study measurements, percentage of successfully completed study measurements. | From enrollment to the end of the study (three months after inclusion)
  Feasibility of study measurements will be assessed by the percentage of successfully completed study measurements and the reported reasons for unsuccessful measurements.

SECONDARY OUTCOMES:
Energy intake (kcal/day) assessed by self-administered 3-day food diary | At the start of the study (directly after inclusion) and three months after inclusion
  Energy intake will be assessed using a self-administered 3-day food diary and calculated as the average daily energy intake in kilocalories using the Evry software.
Protein intake (g/day) assessed by self-administered 3-day food diary | At the start of the study (directly after inclusion) and three months after inclusion
  Protein intake will be assessed using a self-administered 3-day food diary and calculated as the average daily protein intake in grams using the Evry software.
Protein intake (g/kg/day) assessed by self-administered 3-day food diary | At the start of the study (directly after inclusion) and three months after inclusion
  Protein intake relative to body weight will be assessed using a self-administered 3-day food diary and calculated in grams per kilogram per day using the Evry software.
Protein intake (g/kg fat free mass/day) assessed by self-administered 3-day food diary | At the start of the study (directly after inclusion) and three months after inclusion
  Protein intake relative to kg fat free mass will be assessed using a self-administered 3-day food diary and calculated in grams per kilogram fat free mass per day using the Evry software.
Body weight (kg) | At the start of the study (directly after inclusion) and three months after inclusion
  At the start of the study (directly after inclusion) and three months after inclusion
Body height (cm) | At the start of the study (directly after inclusion) and three months after inclusion
  Body height will be measured in centimeters using a stadiometer.
Body mass Index (BMI, kg/m²) | At the start of the study (directly after inclusion) and three months after inclusion
  BMI will be calculated from measured body weight and height and reported in kg/m².
Nutritional status score (PG-SGA, points) | At the start of the study (directly after inclusion) and three months after inclusion
  Nutritional status will be assessed using the Patient-Generated Subjective Global Assessment (PG-SGA) and reported as total points.
Fat mass (kg) assessed by bioelectrical impedance analysis | At the start of the study (directly after inclusion) and three months after inclusion
  Fat mass will be measured using bioelectrical impedance analysis and reported in kilograms.
Fat-free mass (kg) assessed by bioelectrical impedance analysis | At the start of the study (directly after inclusion) and three months after inclusion
  Fat-free mass will be measured using bioelectrical impedance analysis and reported in kilograms.
Muscle thickness of biceps branchii (cm) assessed by ultrasound | At the start of the study (directly after inclusion) and three months after inclusion
  Muscle thickness of the biceps branchii will be measured using ultrasound and reported in centimeters.
Muscle thickness of vastus intermedius (cm) assessed by ultrasound | At the start of the study (directly after inclusion) and three months after inclusion
  Muscle thickness of the vastus intermedius will be measured using ultrasound and reported in centimeters.
Muscle thickness of rectus femoris (cm) assessed by ultrasound | At the start of the study (directly after inclusion) and three months after inclusion
  Muscle thickness of the rectus femoris will be measured using ultrasound and reported in centimeters.
Handgrip strength (kg) assessed by a hand dynamometer | At the start of the study (directly after inclusion) and three months after inclusion
  Handgrip strength will be measured using a hand dynamometer and reported in kilograms.
Physical activity level (minutes/week) assessed by SQUASH questionnaire | At the start of the study (directly after inclusion) and three months after inclusion
  Physical activity will be assessed using the Short Questionnaire to Assess Health-Enhancing Physical Activity (SQUASH) and reported as minutes of activity per week.
Physical performance assessed with Short Physical Performance Battery (SPPB) total score (points) | At the start of the study (directly after inclusion) and three months after inclusion
  Physical performance will be assessed using the Short Physical Performance Battery and reported as total points
Physical performance will be assessed with the Timed Up and Go test (seconds) | At the start of the study (directly after inclusion) and three months after inclusion
  Physical performance will be assessed using the Timed Up and Go test and reported in seconds.
Length of hospital stay (days) | Between enrollment and the end of the study (three months after inclusion)
  Length of hospital stay will be recorded in days from admission to discharge.
Hospital readmissions within 3 months (number) | Between enrollment and the end of the study (three months after inclusion)
  Readmissions will be recorded as the number of hospital readmissions within three months after inclusion.
Complications assessed by type and severity within 3 months | Between enrollment and the end of the study (three months after inclusion)
  Complications occurring within three months after inclusion will be recorded by type (e.g., infection, cardiac event, surgical complication) and severity using PRO-CTCAE Measurement System. Each complication will be reported per patient, and descriptive statistics will be used to summarize the frequency and severity.
Mortality within 3 months (yes/no) | Between enrollment and the end of the study (three months after inclusion)
  Mortality will be recorded as all-cause mortality within three months after inclusion.
Global health status (quality of life) score (0-100) assessed by EORTC QLQ-C30 | At the start of the study (directly after inclusion) and three months after inclusion
  Global health status will be assessed using the EORTC QLQ-C30 questionnaire and reported on a 0-100 scale, with higher scores indicating better global health.
Physical functioning (quality of life) score (0-100) assessed by EORTC QLQ-C30 | At the start of the study (directly after inclusion) and three months after inclusion
  Physical functioning will be assessed using the EORTC QLQ-C30 questionnaire and reported on a 0-100 scale, with higher scores indicating better physical functioning.
Fatigue score (quality of life) score (0-100) assessed by EORTC QLQ-C30 | At the start of the study (directly after inclusion) and three months after inclusion
  Fatigue will be assessed using the EORTC QLQ-C30 questionnaire and reported on a 0-100 scale, with higher scores indicating more fatigue.
Patient satisfaction of the oral nutritonal supplement (ONS) (qualitative) assessed by semi-structured interview | After three months. Or if they stop earlier with the ONS, then directly after they stopped.
  Patient satisfaction with long-term use of ONS will be assessed using semi-structured interviews. Responses will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Maud Reintjes, MSc, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud university medical center, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Yes
Patients will be asked in the informed consent form whether they agree to the possibility that their measurement data may be shared anonymously for future research. If the patient provides consent and the data are relevant to other studies, these anonymized data may be made available to other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: start date: after finishing inclusion. end date: 15 years thereafter
Access Criteria: Other researchers from Radboudumc and Maastricht UMC will have access to the patients' measurement data in an anonymized form. In consultation with the principal investigator/supervisor, the data's relevance to other research will be discussed. Agreements will then be made regarding data sharing. They will only see the study number assigned to each patient and the measurement outcomes. The data cannot be traced back to individual patients.
  Data will be made accessible for other research through the 'DRE' program.

REFERENCES:
- See also: Agreements made in Green Deal 3.0 — https://www.greendealduurzamezorg.nl/files/1-greendeal-samenwerken-aan-duurzame-zorg-c238.pdf
- See also: Sustainable food in hospitals Green Deal — https://www.greendealduurzamezorg.nl/projecten/duurzame-voeding-in-ziekenhuizen-nfu/
- See also: Projects sustainable nutrition in hospitals Green Deal — https://voedingenbeweging.nu/wp-content/uploads/2024/05/Eindverslag-NFU-project-duurzame-voeding-in-ziekenhuizen.pdf

DOCUMENTS (1):
  • Study Protocol (2025-12-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT07399886/Prot_000.pdf